CLINICAL TRIAL: NCT06951503
Title: A Randomized, Controlled, Multicenter Phase III Clinical Study of AK112 Combined With Chemotherapy Versus Bevacizumab Combined With Chemotherapy in First-line Metastatic Colorectal Cancer
Brief Title: A Phase III, Randomized, Controlled and Multi-center Study of AK112 and Chemotherapy in First-line Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK112-312
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Adenocarcinoma
MeSH Terms: interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK112 in combination with FOLFOXIRI (Experimental): AK112 in combination with FOLFOXIRI (Irinotecan, Oxaliplatin, Leucovorin and 5-FU) for induction treatment. Later, patients will receive maintenance Leucovorin and 5-FU plus AK112.
  Interventions: Drug: AK112; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin and 5-FU
- Bevacizumab in combination with FOLFOXIRI (Active Comparator): Bevacizumab in combination with FOLFOXIRI (Irinotecan, Oxaliplatin, Leucovorin and 5-FU) for induction treatment. Later, patients will receive maintenance Leucovorin and 5-FU plus Bevacizumab .
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin and 5-FU; Drug: Bevacizumab

INTERVENTIONS:
Drug: AK112 — iv, q2w
  Arms: AK112 in combination with FOLFOXIRI
Drug: Oxaliplatin — iv, q2w
Drug: Irinotecan — iv, q2w
Drug: Leucovorin and 5-FU — iv, q2w
Drug: Bevacizumab — iv, q2w
  Arms: Bevacizumab in combination with FOLFOXIRI

SUMMARY:
This trial is a Phase III study. The purpose of this study is to evaluate the efficacy and safety of AK112 and chemotherapy versus bevacizumab and chemotherapy for the first-line treatment of metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age ≥ 18 years and ≤ 75 years.
3. ECOG status of 0 or 1.
4. Estimated survival ≥ 3 months.
5. Subjects with histologically or cytologically confirmed metastatic colorectal adenocarcinoma.
6. Subjects who are not candidates for radical surgical resection or local therapy and have not received systemic anti-tumor therapy in the recurrent or metastatic setting. Subjects who have received prior neoadjuvant or adjuvant therapy and whose first discovery of recurrence or metastases is ≥ 12 months after the last dose of neoadjuvant or adjuvant therapy are allowed to enroll.
7. At least one measurable disease based on RECIST v1.1.
8. Adequate organ function per protocol-defined criteria.
9. Women of childbearing potential and men with female partners of childbearing potential must agree to use effective contraception during treatment and for at least 180 days following the last dose of study treatment.

Exclusion Criteria:

1. Previous (within 3 years) or concurrent other malignant tumors, excluding those that have been cured.
2. Participating in other interventional study within 4 weeks prior to the first study drug administration.
3. Palliative local treatment for non-target lesions within 2 weeks prior to the first administration; received non-specific immunomodulatory therapy within 2 weeks prior to the first administration.
4. Current presence of uncontrolled combined disease.
5. Active clinical infections.
6. History of severe bleeding tendency or coagulation dysfunction.
7. Subjects with known active tuberculosis (TB); suspected active TB should be excluded by clinical examination, known active syphilis infection.
8. Received a live vaccine within 30 days prior to the study, or plan to receive a live vaccine during the study.
9. Current presence of significant radiographic or clinical manifestations of GI obstruction.
10. Toxicities of prior anticancer therapy have not resolved to ≤ Grade 1 (NCI-CTCAE version 5.0).
11. Pregnant or lactating women.
12. Any condition considered by the investigator to be inappropriate for enrollment.
13. Local or systemic disease caused by non-malignancy, or disease or symptom secondary to tumor, that can lead to higher medical risk and/or uncertainty in survival.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2025-05-09 (Estimated); Primary Completion 2027-01-13 (Estimated); Study Completion 2029-01-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by blinded independent central review (BICR) | Up to approximately 3 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first (based on RECIST 1.1 criteria).

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization to death due to any cause.
Progression-free survival (PFS) assessed by investigator | Up to approximately 3 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first (based on RECIST 1.1 criteria).
Objective Response Rate (ORR) | Up to approximately 3 years
  ORR is defined as proportion of subjects who have a complete or partial response relative to baseline according to RECIST 1.1 criteria.
Duration of Response (DoR) | Up to approximately 3 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression(based on RECIST v1.1 criteria) or death due to any cause, whichever occurs first.
Disease control rate (DCR) | Up to approximately 3 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (based on RECIST v1.1 criteria).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Sixth Hospital,Sun Yat-sen University, Guanzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided